CLINICAL TRIAL: NCT05075759
Title: SALSA: Study of Active LifeStyle Activation
Brief Title: Testing Counseling and Mobile Health Interventions to Improve Physical Activity and Diet Quality in Survivors of Childhood Cancer
Acronym: SALSA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: RG1121690; NCI-2021-09186 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10784 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA263144 (NIH)
Record Dates: First submitted 2021-09-13; First posted 2021-10-13 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Behavior Therapy; Interviews as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (personalized clinician-led self-management telehealth) (Experimental): Patients receive a personalized clinician-led self-management telehealth session at baseline and 2 months. Patients with poor response at 3 months are randomized to Arm 2 or 4, otherwise patients receive the same telehealth session at months 4 and 6. Patients may receive 2 additional telehealth sessions after 6 months.
  Interventions: Behavioral: Behavioral Intervention; Other: Survey Administration; Other: Interview
- Arm 2 (personalized goal setting) (Experimental): Patients receive personalized goal setting for daily steps and activity (updated weekly) and 3 dietary goals (updated monthly) with social media peer support for 6 months. Patients with poor response at 3 months are randomized to Arms 1 or 4. Patients may receive personalized goal setting for daily steps and activity (updated monthly) and dietary goals (updated monthly) after 6 months.
  Interventions: Behavioral: Behavioral Intervention; Other: Survey Administration; Other: Interview
- Arm 3 (waitlist) (Active Comparator): Patients receive no intervention for 12 months. After 12 months, they may optionally receive their choice of intervention for up to 6 months.
  Interventions: Other: Survey Administration; Other: Interview
- Arm 4 (remote sessions with a health coach) (Experimental): Arm 1 and 2 patients with poor response after 3 months can be re-randomized to Arm 4. Patients receive remote sessions with a health coach every 1-2 weeks for 3 months. Patients may continue to receive remote sessions once a month after 3 months, during the maintenance phase (months 6-12).
  Interventions: Behavioral: Behavioral Intervention; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive personalized clinician-led self-management telehealth sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm 1 (personalized clinician-led self-management telehealth)
Behavioral: Behavioral Intervention — Receive personalized goal setting for daily steps and activity and dietary goals
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm 2 (personalized goal setting)
Behavioral: Behavioral Intervention — Remote sessions with a health coach
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm 4 (remote sessions with a health coach)
Other: Survey Administration — Ancillary studies
Other: Interview — Ancillary studies
  Arms: Arm 1 (personalized clinician-led self-management telehealth); Arm 2 (personalized goal setting); Arm 3 (waitlist)

SUMMARY:
This clinical trial evaluates several behavioral interventions for the improvement of physical activity in cancer patients. Childhood and adolescent/young adult cancer survivors have been reported to have poor diet quality and rarely meet recommended physical activity guidelines. This trial aims to see whether a tailored intervention based on self-determination theory may help to improve physical activity and dietary change.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to Arms 1, 2, or 3.

ARM 1: Patients receive a personalized clinician-led self-management telehealth session at baseline and 2 months. Patients with poor response at 3 months are randomized to Arm 2 or 4, otherwise patients receive the same telehealth session at months 4 and 6. Patients may receive 2 additional telehealth sessions after 6 months.

ARM 2: Patients receive personalized goal setting for daily steps and activity (updated weekly) and 3 dietary goals (updated monthly) with social media peer support for 6 months. Patients with poor response at 3 months are randomized to Arms 1 or 4. Patients may receive personalized goal setting for daily steps and activity (updated monthly) and dietary goals (updated every 2 months) after 6 months.

ARM 3: Patients receive no intervention for 12 months. After 12 months, they may optionally receive their choice of intervention for up to 6 months.

ARM 4: If Arms 1 or 2 patients have poor response after 3 months, patients may be re-randomized to Arm 4. Patients receive remote sessions with a health coach every 1-2 weeks for 3 months. Patients may continue to receive remote sessions once a month after 3 months, during the maintenance phase (months 6-12).

ELIGIBILITY:
Inclusion Criteria:

* Childhood Cancer Survivor Study (CCSS) participant who is between age 18 to < 55 years at time of initial approach
* Moderate to high CV risk status based on CCSS risk prediction models for cardiomyopathy and ischemic heart disease
* Able to read, write, and speak English
* Ability to understand and the willingness to provide informed consent
* At least one of the following:

  * Less than 30 minutes/day of moderate to vigorous physical activity (MVPA) based on validated self-report instrument (Godin)
  * Healthy Eating Index (HEI)-2015 score < 60 per study food frequency questionnaire (FFQ)
  * Body mass index (BMI) >= 25 kg/m^2 per self-reported height and weight
* Be free of any known (self-reported) ischemic heart disease or cardiomyopathy
* Have internet access (can be via smartphone or computer; if neither device is available, the study can loan participants a Wi-Fi enabled device, but participant will need to have access to the internet)

Exclusion Criteria:

* Individuals with known cardiomyopathy or ischemic heart disease based on prior CCSS surveys are excluded. While not likely to be common, participants who newly report in our study's screening questionnaire that they have newly diagnosed cardiomyopathy or ischemic heart disease will also be excluded
* Having any self-reported contraindication to walking or being physically active
* Not currently known to be pregnant; individuals known to be pregnant and otherwise eligible for the study can be enrolled once no longer known to be pregnant. Participants who report being pregnant after randomization can remain in the study
* Individuals receiving active cancer treatment. Participants who report starting active cancer treatment after randomization can remain in the study

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sedentary time | Up to 12 months
  <100 counts/minute as measured by research-grade accelerometry
Healthy Eating Index (HEI)-2015 score | Up to 12 months
  On a scale of 100 (perfect score) as measured by Food Frequency Questionnaire

SECONDARY OUTCOMES:
Participant engagement | Up to 12 months
  As measured by: 1) response to clinician action plans [score of 0-10; 10 being most engaged]; 2) use of mHealth apps [e.g., number of days with daily steps ≥500; number of days with recorded calories ≥500; social media interactions counting viewing, liking, or posting comments]; and 3) number of sessions completed with lifestyle health coach and coach's rating of engagement [score of 0-10; 10 being most engaged]
Health-related self-efficacy scale | Up to 12 months
  Per Schwarzer R, et al. and converted to T-score (higher equaling greater self-efficacy)
Multidimensional Health Locus of Control Scale | Up to 12 months
  Per Wallston KA, et al. with 3 subscales: internal, chance, and powerful others (each scored from 6-36, with higher values indicating greater agreement with that subscale's locus on control beliefs)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Chow, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT05075759/ICF_000.pdf